CLINICAL TRIAL: NCT04948879
Title: A Review of Surgical Outcomes for Patients Undergoing En-bloc Vascular Resection and Reconstruction as Part of Exenteration for Advanced Pelvic Malignancy
Brief Title: The Role of Vascular Reconstruction in the Setting of Pelvic Exenteration
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: St Vincent's University Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Professor Des Winter, Professor Des C Winter, St Vincent's University Hospital, Ireland
Other Study IDs: PelvEx 6
Record Dates: First submitted 2021-06-24; First posted 2021-07-02 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Vascular Reconstruction in Pelvic Exenterative Surgery
MeSH Terms: interventions — Plastic Surgery Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vascular reconstruction: Patients who have undergone resection with or without reconstruction of a major blood vessel in the context of surgery for a locally advanced pelvic malignancy. This will mostly refer to patients who have had resection/reconstruction of their internal iliac vessels, or less likely common iliacs.
  Interventions: Procedure: Vascular resection/reconstruction

INTERVENTIONS:
Procedure: Vascular resection/reconstruction — The resection of a major blood vessel with or without reconstruction

SUMMARY:
Local invasion or abutment of a major vascular structure was once a major deterrent to planned oncological resection. Improvements in radiological assessment and vascular surgical techniques have enabled resection of major blood vessels where focally involved. However, most of this has been conducted in the context of cancers of sarcomatous, hepaticopancreaticobilary or otolaryngological origin, with little evidence detailing the experience in the context of pelvic malignancy. The aim of this retrospective review is to examine the indications for, techniques used and surgical outcomes of vascular reconstruction in the setting of pelvic exenterative surgery.

DETAILED DESCRIPTION:
The role of pelvic exenteration in the management of locally advanced and recurrent pelvic malignancies is ever evolving, with technical advancements enabling surgeons to perform more radical resections, offering a potential cure to many patients who would have once been deemed inoperable. As surgical oncology has shifted towards higher-volume, specialist centres in a bid to improve outcomes, surgeons have used greater experience to re-evaluate what can be considered as resectable disease. This is best exemplified by a trend towards en bloc vascular excision and reconstruction where tumours abut or focally invade adjacent vasculature. Whereas involvement of a major vascular structure remains a relative contraindication to surgery in some units (1), certain specialist centres around the world are increasingly reporting on the feasibility of this approach.

It is accepted that achieving an R0 resection is the most significant prognostic factor for overall survival (OS) in exenterative surgery. Conversely, involvement of the lateral compartment is a poor prognostic variable, in large part due to the difficulty obtaining a negative resection margin without compromising neurovascular structures(2). Improvements in pre-operative radiological assessment, particularly with respect to angiography, have facilitated appropriate patient and treatment selection, while advancements in the field of vascular surgery have made the procedure technically feasible.

However, there is no clear consensus on the role of vascular reconstruction in curative treatment of advanced pelvic malignancy, owing to a paucity of published data. Initial reports and series have shown promising results, but these are almost exclusively single-surgeon experiences with small numbers and heterogenous populations. Therefore, there is a need for collaborative data to assess the impact and success of such surgical strategies.

The aim of this retrospective review is to examine the indications for, techniques used and surgical outcomes of vascular reconstruction in the setting of pelvic exenterative surgery at a multicentre level in order to inform future practice, with a particular focus on whether or not it significantly increases the morbidity in the short-term.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven locally advanced or recurrent pelvic cancer (all subtypes, RECTAL, UROLOGICAL, GYNAE, SARCOMA)
* Aged over 18 years
* Undergoing a multi-visceral extended pelvic resection
* Requiring a vascular resection with or without the need for reconstruction as part of pelvic exenteration

Exclusion Criteria:

* Strong evidence of metastatic or peritoneal disease
* No histological evidence of vascular structures resected at time of operation
* Insufficient patient follow-up (Minimum of 30 days)
* Insufficient information on post-operative follow-up of graft patency/function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 years who undergo resection/reconstruction of a major blood vessel as part of pelvic exenteration for a locally advanced or recurrent pelvic (rectal, urological, gynaecological, sarcomatous) malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Morbidity | July 2016 - July 2021
  Post-operative complications (<30 days), as measured by the Clavien-Dindo scale

SECONDARY OUTCOMES:
Blood loss | July 2016 - July 2021
  Blood loss (mL)
Length of stay | July 2016 - July 2021
  Duration of stay in hospital post-procedure
Graft patency/function | July 2016 - July 2021
  Whether or not the reconstruction is functioning
Resection status | July 2016 - July 2021
  Resection margins (R0, R1 or R2)
Mortality | July 2016 - July 2021
  Proportion of patients who die within 30 days of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Winter, MD, Study Chair — St. Vincent's Healthcare Group

IPD SHARING:
Plan to Share IPD: No
Patient data will be anonymised by participating PelvEx centres and then shared with the collaborative.